CLINICAL TRIAL: NCT04224337
Title: Phase II Study of Durvalumab ,Doxorubicin, and Ifosfamide in Pulmonary Sarcomatoid Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Bhumsuk Keam, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSC2
Record Dates: First submitted 2020-01-08; First posted 2020-01-13 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Doxorubicin; Ifosfamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Durvalumab + doxorubicin + ifosfamide
  Interventions: Drug: Durvalumab + doxorubicin + ifosfamide

INTERVENTIONS:
Drug: Durvalumab + doxorubicin + ifosfamide — Durvalumab: 1500mg via IV infusion on day 1 Q3W for 4 cycles followed by durvalumab monotherapy 1500mg via IV infusion Q4W for up to a maximum 12 months Doxorubicin 20mg/m2 via IV infusion on day 1 to day 3 Q3W (up to 4 cycles) Ifosfamide: 1.5g/m2 (with mesna) via IV infusion on day 2 to day 4 Q3W (up to 4cycles)

SUMMARY:
To evaluate the efficacy and safety of durvalumab in combination with doxorubicin and ifosfamide in patients with PSC.

DETAILED DESCRIPTION:
This is a phase II multi-center, open-label study to evaluate the efficacy and safety of durvalumab in combination with doxorubicin and ifosfamide in patients with PSC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed NSCLC with the histology of sarcomatoid carcinoma (WHO criteria for sarcomatoid carcinoma is used; carcinoma with spindle and/or giant cells, pleomorphic carcinoma, spindle cell carcinoma, giant cell carcinoma, carcinosarcoma, pulmonary blastoma). If the NSCLC patients showed sarcomatoid carcinoma histology in re-biopsy sample (so called epithelial-mesenchymal transition (EMT) phenomenon), such patients are eligible.
2. Age ≥ 20 years at time of study entry.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Initial metastatic cases or recurrent cases after curative treatment (up to 2 previous lines are allowed, and patients who experienced immune-checkpoint inhibitors are also allowed).
5. A patient with at least one measurable lesion by RECIST1.1.
6. Asymptomatic brain metastasis. If patients have brain metastasis with neurological symptom, they should be stabilized neurologically with prior radiotherapy or surgery for the brain metastasis.
7. Body weight >40kg
8. Adequate normal organ and marrow function as defined below:

   * Haemoglobin ≥9.0 g/dL
   * Absolute neutrophil count (ANC) ≥ 1,500 /mm3
   * Platelet count ≥100,000 /mm3
   * Serum bilirubin ≤1.5 x upper limit of normal (ULN).
   * AST (SGOT)/ALT (SGPT) ≤2.5 x ULN unless liver metastases are present, in which case it must be ≤5x ULN
   * Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976)
9. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

   Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy). Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
10. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
11. Must have a life expectancy of at least 12 weeks.
12. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 3weeks.
2. A patient with no measurable disease.
3. History of diverticulitis, intra-abdominal abscess, gastrointestinal obstruction, abdominal carcinomatosis which are known risks factors for bowel perforation.
4. Active autoimmune disease within the past 2 years (NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment -within the past 2 years- are not excluded) or a documented history of autoimmune disease or syndrome that requires systemic steroids or immunosuppressive agents.
5. Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤ 3 weeks prior to the first dose of study drug If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period will be required, as agreed by AstraZeneca/MedImmune and the investigator.
6. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
7. Any concurrent chemotherapy, IP, or biologic therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
8. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
9. History of allogenic organ transplantation.
10. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid.
11. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    3. Any chronic skin condition that does not require systemic therapy
    4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    5. Patients with celiac disease controlled by diet alone
12. Uncontrolled current illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
13. History of another primary malignancy except for

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    3. Adequately treated carcinoma in situ without evidence of disease, NED ≥3 years
14. History of cytologically proven leptomeningeal carcinomatosis
15. QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECG
16. A patient with clinically significant (i.e. active) heart disease (e.g.congestive heart failure, symptomatic coronary artery diseases, cardiac arrhythmias, etc) or myocardial infarction within past 12 months.
17. History of active primary immunodeficiency.
18. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) and with appropriate prophylactic antiviral agents for positive HbsAg are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
19. Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
20. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
21. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of durvalumab monotherapy.
22. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
23. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Response rate (RR) | 24 months
  modified RECIST1.1, a percentage and is calculated by dividing the number of patients who achieved a response (complete or partial) by the total number of evaluable patients in the study

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 24 months
  the percentage of patients who have not experienced disease progression or death from any cause within 2 years from the start of treatment.
Overall survival (OS) | 24 months
  The duration of time from the start of treatment until death from any cause
Adverse event | 24 months
  The number of patients with treatment-related AE as assessed by NCI CTCAE

OTHER OUTCOMES:
biomarker | 24 months
  Correlation with C-MET mutation, PD-L1 IHC

CONTACTS AND LOCATIONS:
Overall Officials: Bhumsuk Keam, Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
anticipated as research paper